CLINICAL TRIAL: NCT05982080
Title: A Phase 1 Study to Investigate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics Activity of FP002 in Subjects With Advanced Malignancies
Brief Title: A Study to Investigate FP002 in Subjects With Advanced Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Fapon Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP002-CT1001-CN
Record Dates: First submitted 2023-07-07; First posted 2023-08-08 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FP002 Injection (Experimental): Dose escalation: FP002
  Interventions: Drug: FP002 Injection

INTERVENTIONS:
Drug: FP002 Injection — Up to 6 FP002 dose levels (0.3, 1.0, 3.0, 10, 20, 30 mg/kg administered intravenously may be evaluated. Subjects will receive weekly infusions of FP002 until disease progression, unacceptable toxicity, consent withdrawal, physician decision, or start of subsequent anticancer therapy, whichever occurs first.

SUMMARY:
The goal of this phase 1 study is to assess the safety, and tolerability of FP002 to determine the dose recommended for dose expansion in subjects with advanced solid tumor.

DETAILED DESCRIPTION:
This study is a phase 1 study of FP002 as monotherapy in patients with advanced solid tumor. The study will evaluate the safety, tolerability, pharmacokinetic, pharmacodynamic profile, immunogenicity, and preliminary anti-tumor activity of FP002 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF) and was able to comply with the protocol.
2. Male or female subjects ≥ 18 years of age on the day of ICF signing.
3. A life expectancy of > 3 months.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Adequate organ and bone marrow function confirmed at screening and within 7 days before the first dose of study treatment.
6. Subjects with histologically or cytological confirmed malignancy diagnosis.
7. Documented advanced solid tumors, defined as patients have no standard treatment or who have failed/are intolerant to standard treatment according to the investigator's judgment.
8. Documented with at least 1 measurable lesion as assessed by RECIST 1.1.
9. Toxicity from prior anti-tumor treatment has resolved to ≤ Grade 1 as defined by NCI CTCAE v5.0.

Exclusion Criteria:

1. Subjects who have received other anti-CD47 or anti- SIRPα agents.
2. Prior organ or tissue allograft except for hematopoietic stem cell transplantation.
3. Treatment with investigational therapy within 4 weeks prior to initiation of study drug.
4. Severe infection requiring hospitalization or IV antibiotics, antivirals or antifungals within 14 days prior to enrollment.
5. Subjects who have received chemotherapy within 4 weeks or 5 half-lives (whichever is shorter) before the first dose (within 6 weeks before the first dose of mitomycin or nitrosoureas) or received immunotherapy, radical radiotherapy or major surgery within 4 weeks or palliative radiotherapy within 2 weeks.
6. Subjects who have experienced active autoimmune disease requiring systemic therapy within the past 2 years.
7. A positive test result for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by a certified nucleic acid test within the last 30 days before the first dose of study treatment.
8. Cardiovascular dysfunction or clinically significant cardiac disease.
9. Active infection with hepatitis C.
10. Receipt of a live vaccine within 30 days prior to the first dose of study treatment.
11. Known hypersensitivity to either the drug substances or inactive ingredient of FP002.
12. Known human immunodeficiency virus (HIV) positive.
13. A history of other malignancies other than effectively treated basal cell carcinoma of skin, squamous cell carcinoma of skin, or effectively resected carcinoma in situ of the cervix.
14. Known inherited or acquired bleeding disorders.
15. Any other medical, family, social or mental conditions that the investigator considers unsuitable for participation in the study.
16. Daily requirement for corticosteroids (≥10 mg/kg) within 2 weeks prior to Day 1 of Cycle 1.
17. Women who are lactating or pregnant as confirmed by pregnancy test within 7 days before the first dose of study treatment. Unwilling to use adequate contraceptive methods during the study and for at least 7 months after the last dose of study treatment.
18. Presence of active brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Severity (as graded by CTCAE v5.0) of Dose Limiting Toxicity (DLT) | During the first 4 week treatment cycle
Severity (as graded by CTCAE v5.0) of treatment-emergent AEs (TEAEs) | up to 24 months
Severity (as graded by CTCAE v5.0) of serious adverse events (SAEs) | up to 24 months
Severity (as graded by CTCAE v5.0) of adverse events of special interest (AESIs) | up to 24 months
Severity (as graded by CTCAE v5.0) of adverse events assessed | up to 24 months

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of FP002 | up to 24 months
Area under the curve from time zero to the last measurable time point (AUC0-t) of FP002 | up to 24 months
Area under the curve extrapolated to infinity (AUC0-inf)of FP002 | up to 24 months
Time to reach maximum plasma concentration (Tmax) of FP002 | up to 24 months
Terminal elimination half-life (t1/2) of FP002 | up to 24 months
Apparent volume of distribution (Vd) of FP002 | up to 24 months
Clearance rate (CLz) | up to 24 months
Terminal elimination rate constant (λz) | up to 24 months
Mean retention time (MRT) | up to 24 months
Maximum plasma concentration during the dosing interval at steady state (Cmax,ss) | up to 24 months
Minimum plasma concentration during the dosing interval at steady state (Cmin,ss) | up to 24 months
Average steady state concentration (Cav) | up to 24 months
Steady-state clearance rate (CLss) | up to 24 months
Steady-state volume of distribution (Vss) | up to 24 months
Accumulation index (Rac) | up to 24 months
Degree of fluctuation (DF) | up to 24 months
Duration of response (DoR) based on RECIST V1.1 | Up to 24 months
Disease control rate (DCR) based on RECIST V1.1 | Up to 24 months
Overall response rate (ORR) based on RECIST V1.1 | Up to 24 months
Progression free survival (PFS) based on RECIST V1.1 | Up to 24 months
Anti-drug antibody | Up to 24 months
  Incidence, onset time and titer
Neutralizing antibody | Up to 24 months
  Incidence, onset time and titer
Receptor of occupancy in RBC/CD3+ T cell | Up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Yuping Sun, MD, Principal Investigator — Shangdong Cancer Hospital & Institute; Linlin Wang, MD, Principal Investigator — Shangdong Cancer Hospital & Institute
Locations (3):
- China (3):
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Shangdong Cancer Hospital & Institute, Jinan, Shangdong
  - Linyi Cancer Hospital, Linyi, Shangdong

IPD SHARING:
Plan to Share IPD: No